CLINICAL TRIAL: NCT06572085
Title: Neuroprotective Effect of Butylphthalide Injection on Patients With Return of Spontaneous Circulation After Cardiac Arrest：a Multicenter, Randomized Clinical Trial
Brief Title: Neuroprotective Effect of Butylphthalide for Cardiac Arrest Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tang Ziren (Other)
Responsible Party: Sponsor-Investigator, Tang Ziren, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-11-30-4
Record Dates: First submitted 2024-08-25; First posted 2024-08-26 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Butylphthalide; Cardiac Arrest; Neuroprotective Drugs
MeSH Terms: conditions — Heart Arrest | interventions — 3-n-butylphthalide; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Butylphthalide (Experimental): Butylphthalide and Sodium Chloride Injection 100ml ivgtt bid 14days
  Interventions: Drug: Butylphthalide and Sodium Chloride Injection
- Saline Solution (Placebo Comparator): Saline Solution 100ml ivgtt bid 14days
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Butylphthalide and Sodium Chloride Injection — All enrolled patients will undergo standard treatment as per international guidelines, concurrently receiving either NBP or placebo therapy. Patients in the experimental group will receive intravenous infusion of 100ml NBP injection twice daily, while patients in the control group will receive intravenous infusion of 100ml saline solution twice daily. Each patient will receive continuous medication for 14 days.
  Arms: Butylphthalide
Drug: Saline Solution — All enrolled patients will undergo standard treatment as per international guidelines, concurrently receiving either NBP or placebo therapy. Patients in the experimental group will receive intravenous infusion of 100ml NBP injection twice daily, while patients in the control group will receive intravenous infusion of 100ml saline solution twice daily. Each patient will receive continuous medication for 14 days.
  Arms: Saline Solution

SUMMARY:
Cardiac arrest is one of the critical illnesses that is directly life-threatening, and patients who survive cardiac arrest develop severe neurological deficits or even die. The effectiveness of drugs to improve neurological function in resuscitated brain-injured patients has been a focus of research in the field of resuscitation. Butanephthalein has an ameliorating effect on the damage of central nervous function in patients with acute ischemic stroke, and can promote the improvement of patients' neurological deficits. On this basis, the present study was designed as a multicenter, prospective randomized controlled experiment, with internationally accepted methods for assessing near-term and long-term neurological function, to determine the effectiveness of butalbital in improving neurological function after cardiac arrest, with the aim of searching for new methods and ideas to improve neurological function and prognosis after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old.
2. Glasgow Coma Scale (GCS) scores ≤8 upon admission.
3. Return of Spontaneous Circulation (ROSC) ≥30min.
4. Signed the informed consent form.

Exclusion Criteria:

1. Cardiac arrest due to irreversible causes such as trauma, poisoning, etc.
2. Cardiac arrest due to end-stage conditions such as advanced cancer.
3. Persistent cardiogenic shock that is unreversed (defined as a systolic blood pressure persistently <90mmHg despite treatment with fluid resuscitation, vasopressor agents, and inotropic medications).
4. Presence of pre-existing cerebrovascular disease prior to cardiac arrest or confirmed intracranial hemorrhage by CT scan following admission.
5. Pre-existing CPC scores of 3-5 prior to cardiac arrest.
6. Prior use of NBP or any medication containing NBP before cardiac arrest.
7. Presence of severe hepatic or renal dysfunction before cardiac arrest (defined as ≥3× upper limit of normal alanine transaminase or ≥2× upper limit of normal creatinine).
8. Bradycardia or sick sinus syndrome occurs after ROSC.
9. History of prior drug or food allergies, or known allergies to the medication components used in this study.
10. Existence of treatment limitations (patient or their legal representative refusing advanced life support treatment, including mechanical ventilation, chest compressions, targeted temperature management, etc.).
11. Presence of severe bleeding tendency upon admission.
12. Body temperature <30℃ upon admission.
13. Pregnant or lactating women, or reproductive-age females with elevated serum human Chorionic Gonadotropin (hCG) levels.
14. Other conditions deemed unsuitable for this trial by the principal investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a Cerebral Performance Category (CPC) Score of 1-2 | 6 months
  The primary outcome is the proportion of patients with a Cerebral Performance Category (CPC) score of 1-2 at 6months after randomization in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chao-Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: The de-identified survey data will be made available for research purposes by contacting the corresponding authors